CLINICAL TRIAL: NCT01685606
Title: BrUOG 273:Cellular Immunotherapy For Refractory Hematological Malignancies:A Brown University Oncology Research Group Study
Brief Title: Study of Infusion of Blood Cells (Lymphocytes) to Stimulate the Immune System to Fight Leukemia/Lymphoma
Acronym: 273
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual and low efficacy
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 273
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Mantle Cell Lymphoma; Diffuse Large Cell Lymphoma; Burkitts Lymphoma; T Cell Lymphomas; Acute Myeloid Leukemia/Acute Lymphoblastic Leukemia
Keywords: Leukemia; Lymphoma; Mantle cell; DLBCL; DLBC; Diffuse large B cell; T cell; AML; ALL
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, T-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cellular immunotherapy (Experimental): A minimum of 1x108 CD3+ cells and maximum of 2x108 CD3+ cells/kg from a haploidentical donor will be infused, irrespective of the number of CD34+ cells.
  Interventions: Biological: cellular immunotherapy

INTERVENTIONS:
Biological: cellular immunotherapy — A minimum of 1x108 CD3+ cells and maximum of 2x108 CD3+ cells/kg from a haploidentical donor irrespective of the number of CD34+ cells will be infused.

SUMMARY:
The study of whether an infusion of blood cells called lymphocytes from a donor can stimulate the immune system to fight your leukemia/lymphoma.

DETAILED DESCRIPTION:
There have been important advances in the modulation of the immune system for the treatment of hematologic malignancies and solid tumors.

This protocol will build upon these previous observations as follows:

* Haploidentical peripheral blood pheresed cells will be used at 1-2x108 CD3 cells/kg.
* Total body radiation will not be utilized.

  * This modification may more effectively activate the recipient's immune system to attack their hematological malignancy by not damaging the recipient's immune cells prior to cellular infusion. Safety should be improved since the risk of graft versus host disease should be greatly reduced as the host's immune system will not be conditioned.
* Granulocyte-colony stimulating factor (G-CSF) priming will not be used.

  * In our first clinical trial, G-CSF priming was not used for matched transplants. Our second trial did employ G-CSF priming in the haplo-identical setting. Previous data has cited a role for G-CSF in stimulation of invariant Natural Killer(NK) cells with enhanced GVL effects11. However, our most recent laboratory data with unprimed PBMC has shown effective cell kill activity without the addition of G-CSF. As G-CSF would be administered to healthy volunteers, the unclear benefit of the addition of this cytokine is offset by the potential side effects such as headache, fever, and bone pain. G-CSF mobilization serves to shift the response from a TH1 to TH2 through the increased production of T regulatory cells. The end result would be a decrease in immune stimulation. Since the goal of this study is to NOT have engraftment, the manipulation of the donor cells to dampen the host versus tumor stimulation is not needed nor desired. Furthermore, since this protocol is not a stem cell transplant, stem cells do not need to be mobilized with G-CSF.

It is important to note that the proposed study is not a stem cell transplant study. In the situation of stem cell transplants, the goal of the procedure is to have engraftment, or sustainable donor chimerism in the marrow to provide hematopoietic reconstitution as well as immunologic reconstitution. In this study, we are evaluating the use of donor lymphocytes (not stem cells) to stimulate an immune response of the recipients' immune system.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of hematological malignancy consisting of the following leukemias/lymphomas:
* Mantle cell lymphoma with Ki-67>30%
* Diffuse Large Cell Lymphoma
* Burkitts Lymphoma
* Systemic T Cell Lymphomas
* Acute Myeloid Leukemia
* Acute Lymphoblastic Leukemia
* Recurrence or progression of hematological malignancy after at least 1 prior standard treatment with progression within 6 months from last treatment.
* No curative treatment option is available.

  -> 4-weeks since prior chemotherapy or radiation to cellular therapy infusion. (Hydroxyurea may be utilized up to 48 hours prior to initiation of treatment on this protocol).
* Age equal to or greater than 18 years.
* Patients with a history of invasive second malignancy unless disease free for > 5 years.
* Patients must have an expected life expectancy of at least 2 months at the time of initiation of treatment.
* No active systemic infection.
* Patients who have relapsed after standard autologous stem cell infusion are eligible as long as they meet all inclusion criteria and no exclusion criteria. These patients must be out more than 6 months from cell infusion to be eligible for enrollment.
* DLCO > 40% with no symptomatic pulmonary disease.
* LVEF > 40% by MUGA or echocardiogram.
* Creatinine < 2.0 mg/dl. Total bilirubin less than 1.5x the upper limit of normal (ULN), AST < 3x ULN.
* Non-pregnant and willing to use appropriate birth control during the duration of the study period.

Exclusion Criteria:

* Evidence of HIV infection.
* Any uncontrolled severe, concurrent illness which in the opinion of the treating physician would make this protocol treatment unreasonably hazardous for the patient.
* Oxygen dependent obstructive pulmonary disease.
* Failure to demonstrate adequate compliance with medical therapy and follow-up.
* Significant medical or psychiatric illness that would impair the ability to participate in protocol therapy.
* For women of reproductive potential, refusal to use effective form of contraception.
* Previous allogeneic stem cell transplant
* Patients who have had previous purine analog (fludarabine, pentostatin, 2-CDA) -Patients with chronic myeloid leukemia (CML), chronic lymphocytic leukemia (CLL), multiple myeloma, and indolent lymphoma (follicular lymphoma, marginal zone lymphoma)
* Patients with HLA antibodies to donor HLA type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Quesenberry, MD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Reagan JL, Fast LD, Safran H, Nevola M, Winer ES, Castillo JJ, Butera JN, Quesenberry MI, Young CT, Quesenberry PJ. Cellular immunotherapy for refractory hematological malignancies. J Transl Med. 2013 Jun 19;11:150. doi: 10.1186/1479-5876-11-150. PMID 23782682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cellular Immunotherapy
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cellular Immunotherapy
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 66.2 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Cellular Immune Therapy With HLA Haploidentical Peripheral Blood Pheresed Cells in Patients With Relapsed/Refractory Hematological Malignancies.
Description: Criteria for AML and ALL (adapted from Cheson et al.20)
  Complete remission (CR) is defined as the presence of all of the following
  * Peripheral blood
    o No leukemic blasts present.
  * No extramedullary findings of leukemia or disappearance of such (i.e. CNS or soft tissue involvement)
  * Bone marrow
    * Cellularity >20% with baseline maturation.
    * No Auer rods
    * Less than 5% blast cells.
  * Complete blood counts and bone marrow normalization criteria must be met within one week of each other. Hematopoeitic recovery is an ANC > 1.0 x 109/L and platelet count > 100x109/L. No specific hemoglobin or hematocrit level is specified but the patient must be transfusion free.
  Complete remission with incomplete recovery (CRi) is defined as the following:
  * Meets criteria for CR except
  * ANC < 1.0 x 109/L or platelet count < 100x109/L
  Partial remission (PR).
  • Must meet all criteria of a CR except that the bone marrow may contain 5-20% blasts.
Time Frame: 8 weeks after infusion then 6 months after and every 4 months for approximately 2 years
Measure: Number; unit: participants
Arm/Group | Cellular Immunotherapy
Number analyzed (Participants) | 5
participants | 1

2. Secondary Outcome: To Evaluate the Rate of Dose Limiting Toxicities of HLA Haploidentical Peripheral Blood Pheresed Cellular Infusions.
Time Frame: 30 days and 16 weeks after infusion
Measure: Number; unit: participants
Arm/Group | Cellular Immunotherapy
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Arm/Group | Cellular Immunotherapy
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellular Immunotherapy (N=6)
Albumin (Investigations) | 1 (1)
ALT (Investigations) | 1 (1)
anemia (Investigations) | 2 (2)
AST (Investigations) | 1 (1)
bone pain (Investigations) | 1 (1)
ca (Investigations) | 1 (1)
CRS (pt 3 included n, ha, r) (Investigations) | 1 (1)
diarrhea (Investigations) | 1 (1)
dizziness (Investigations) | 4 (4)
Febrile Neutropenia (Investigations) | 1 (1)
fever (Investigations) | 2 (2)
Hypotension (Investigations) | 3 (3)
tachycardia (Investigations) | 1 (1)
infection (Investigations) | 1 (1)
(Investigations) | 1 (1)
Nausea (Investigations) | 1 (1)
Neutropenia (Investigations) | 1 (1)
pain-neck (Investigations) | 1 (1)
PLT (Investigations) | 1 (1)
creatinine (Investigations) | 1 (1)
infection: wound (Investigations) | 1 (2)
GI bleed (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellular Immunotherapy (N=6)
alk phos (Investigations) | 1 (1)
anemia (Investigations) | 4 (4)
anxiety (Investigations) | 1 (1)
arthralgia (Investigations) | 1 (1)
bleeding scrotum (Investigations) | 1 (1)
bone pain (Investigations) | 1 (1)
ca (Investigations) | 2 (2)
diarrhea (Investigations) | 1 (1)
cough (Investigations) | 2 (2)
edema (Investigations) | 2 (2)
epistaxis (Investigations) | 1 (1)
erythema (Investigations) | 1 (1)
eye stye Not graded pt 3 (Investigations) | 2 (2)
fever (Investigations) | 2 (2)
Hyperglycemia (Investigations) | 5 (5)
K (Investigations) | 1 (1)
Leukocytosis (Investigations) | 1 (1)
Lymph (Investigations) | 4 (4)
minor bleeding superficila leg lesions "minor" NG pt #3 (Investigations) | 1 (1)
(Investigations) | 2 (2)
Neutropenia (Investigations) | 3 (3)
oral thrush (Investigations) | 1 (1)
Phos (Investigations) | 2 (2)
PLT (Investigations) | 1 (1)
post nasal (Investigations) | 1 (1)
segs/neuts (Investigations) | 1 (1)
sinus pain Not graded pt 3 (Investigations) | 1 (1)
sinus tach (Investigations) | 1 (1)
Vomiting (Investigations) | 1 (1)
WBC (Investigations) | 2 (2)
cellulitis (Investigations) | 1 (1)
fatigue (Investigations) | 1 (1)
LE pain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No